CLINICAL TRIAL: NCT04466436
Title: Effect of Anaesthesia on Tryptophan Pathway
Brief Title: Anaesthesia and Tryptophan Pathway
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rasha Hamed, lecturer of anaesthesia, Assiut University
Other Study IDs: 13700421
Record Dates: First submitted 2020-07-08; First posted 2020-07-10 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Tryptophan Pathway
MeSH Terms: interventions — Tryptophan

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CABG group
  Interventions: Other: tryptophan
- spine group
  Interventions: Other: tryptophan

INTERVENTIONS:
Other: tryptophan — measurement of tryptophan in serum

SUMMARY:
Surgery has many immunomodulatory properties of which the mechanism is not clearly understood.

DETAILED DESCRIPTION:
surgery and anesthesia have a deleterious effect on immune system,studyingtryptophan pathway might give more information on their effect.

ELIGIBILITY:
Inclusion Criteria:

* elective surgery

Exclusion Criteria:

* emergency surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: adults undergoing elective surgery
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2020-07-08 (Actual); Primary Completion 2020-08-08 (Estimated); Study Completion 2020-08-10 (Estimated)

PRIMARY OUTCOMES:
tryptophan metabolites in serum | 72 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt